CLINICAL TRIAL: NCT01412983
Title: A Study to Evaluate the Product Feasibility of a New Silicone Hydrogel Contact Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Screening
Other Study IDs: 713E
Record Dates: First submitted 2011-08-08; First posted 2011-08-09 (Estimated); Results first posted 2014-04-29 (Estimated); Last update posted 2014-04-29 (Estimated); Status verified 2014-03

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bausch & Lomb Test Lens (Experimental): Bausch + Lomb investigational soft contact lens
  Interventions: Device: Bausch & Lomb Test lens
- Ciba Vision soft contact lens (Active Comparator): Ciba Vision Air Optix Aqua soft contact lens
  Interventions: Device: Ciba Vision soft contact lens

INTERVENTIONS:
Device: Bausch & Lomb Test lens — Lens to be worn on a daily wear basis for one week. Participants will be provided with Bausch + Lomb renu® fresh™ multi-purpose solution for daily rinsing, cleaning, and disinfecting of their lenses.
  Arms: Bausch & Lomb Test Lens
Device: Ciba Vision soft contact lens — Lens to be worn on a daily wear basis for one week. Participants will be provided with Bausch + Lomb renu® fresh™ multi-purpose solution for daily rinsing, cleaning, and disinfecting of their lenses.
  Arms: Ciba Vision soft contact lens

SUMMARY:
The objective of this study is to determine the clinical feasibility and to evaluate the product performance of investigational contact lenses developed by Bausch + Lomb.

ELIGIBILITY:
Inclusion Criteria:

* Have physiologically normal anterior segments not exhibiting clinically significant biomicroscopy findings (greater than grade 1 and/or presence of infiltrates).
* Be adapted wearers of soft contact lenses, wear a lens in each eye, and each lens must be of the same manufacture and brand.
* Be correctable through spherocylindrical refraction to 32 letters (0.3 logMAR) or better (distance, high contrast) in each eye.
* Be myopic and require lens correction from -0.50 to -6.00 diopters (D) in each eye.

Exclusion Criteria:

* An active ocular disease, any corneal infiltrative response or are using any ocular medications.
* Have worn gas permeable (GP) contact lenses within last 30 days or PMMA lenses within last 3 months.
* Any Grade 2 or greater finding during the slit lamp examination that, in the Investigator's judgment, interferes with contact lens wear.
* Any scar or neovascularization within the central 4mm of the cornea.
* Have had any corneal surgery.
* Any "Present" finding during the slit lamp examination that, in the Investigator's judgment, interferes with contact lens wear.
* Any systemic disease affecting ocular health.
* Using any systemic or topical medications that will affect ocular physiology or lens performance.
* Currently wear monovision, multifocal, or toric contact lenses.
* Allergic to any component in the study care products.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-08; Primary Completion 2011-09 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Beverly J Barna, CCRA, Study Director — Bausch & Lomb Incorporated
Locations (1):
- Bausch & Lomb Incorporated, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 5 clinical sites in the US. First participant was enrolled 08/08/2011 and last participant exited on 09/01/2011.
Pre-assignment Details: 100 participants (200 eyes) were enrolled in this 2 week crossover study. Participants were divided into 2 groups wearing one study lens for 1 week and then crossing over to the other study lens for 1 week. 96 participants completed the study, 1 participant was ineligible at baseline while 3 participants were discontinued during the study.
Groups:
- Bausch+Lomb Test Lens Then Ciba Vision Lens: Bausch+Lomb investigational soft contact lens
  Bausch+Lomb Test lens:Ciba Vision Lens. Lens to be worn on a daily wear basis for one week. Participants will be provided with Bausch + Lomb renu® fresh™ multi-purpose solution for daily rinsing, cleaning, and disinfecting of their lenses.
- Ciba Vision Soft Contact Lens Then Bausch+Lomb Test Lens: Ciba Vision Air Optix Aqua soft contact lens
  Ciba Vision lens:Bausch+Lomb Test Lens. Lens to be worn on a daily wear basis for one week. Participants will be provided with Bausch + Lomb renu® fresh™ multi-purpose solution for daily rinsing, cleaning, and disinfecting of their lenses.
Period: 1st Period
Arm/Group | Bausch+Lomb Test Lens Then Ciba Vision Lens | Ciba Vision Soft Contact Lens Then Bausch+Lomb Test Lens
Started | 50 | 50
Completed | 50 | 46
Not Completed | 0 | 4
Not completed — Ineligible | 0 | 1
Not completed — Positive slit lamp finding | 0 | 1
Not completed — Unacceptable lens movement | 0 | 1
Not completed — Inability to maintain wear | 0 | 1
Period: 2nd Period
Arm/Group | Bausch+Lomb Test Lens Then Ciba Vision Lens | Ciba Vision Soft Contact Lens Then Bausch+Lomb Test Lens
Started | 50 | 46
Completed | 50 | 46
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants enrolled in the study
Groups:
- Overall Study: All 99 participants in study
Arm/Group | Overall Study
Number analyzed (Participants) | 99
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.9 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67
  Male | 32
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 94
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 99

OUTCOME MEASURES:

1. Primary Outcome: Visual Acuity
Description: The mean difference in high contrast logMAR, over all lens visual acuities (VAs) between lens groups.
Time Frame: One week
Population: All eligible dispensed eyes
Measure: Least Squares Mean (Standard Deviation); unit: LogMAR
Units Other Than Participants: eyes
Groups:
- Bausch+Lomb Test Lens: Bausch+Lomb investigational soft contact lens
  Bausch+Lomb Test lens: Lens to be worn on a daily wear basis for one week. Participants will be provided with Bausch+Lomb renu® fresh™ multi-purpose solution for daily rinsing, cleaning, and disinfecting of their lenses.
Arm/Group | Bausch+Lomb Test Lens | Ciba Vision Soft Contact Lens
Number analyzed (Participants) | 96 | 95
Number analyzed (eyes) | 192 | 190
LogMAR | -0.054 (0.115) | -0.051 (0.115)

2. Secondary Outcome: Overall Comfort
Description: The mean difference in comfort-related symptoms/complaints scores between lens groups. Rated on a scale of 0-100 with 100 being the most favorable score.
Time Frame: One week
Population: All eligible dispensed eyes
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Groups:
- Bausch + Lomb Test Lens: Bausch + Lomb investigational soft contact lens
  Bausch + Lomb Test lens: Lens to be worn on a daily wear basis for one week. Participants will be provided with Bausch + Lomb renu® fresh™ multi-purpose solution for daily rinsing, cleaning, and disinfecting of their lenses.
Arm/Group | Bausch + Lomb Test Lens | Ciba Vision Soft Contact Lens
Number analyzed (Participants) | 96 | 97
Number analyzed (Eyes) | 192 | 194
units on a scale | 81.9 (21.7) | 82.7 (21.8)

ADVERSE EVENTS:
Time Frame: 1 week
Arm/Group | Bausch & Lomb Test Lens | Ciba Vision Soft Contact Lens
Serious Adverse Events (participants affected / at risk) | 0/99 | 0/99
Other Adverse Events (participants affected / at risk) | 0/99 | 0/99

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other